CLINICAL TRIAL: NCT03891394
Title: Prognostic Value of Human Epididymis Protein 4 (HE4) for Persistent Proteinuria in Women With Severe Preeclampsia / HELLP Syndrome
Brief Title: Human Epididymis Protein 4 in Women With Severe Preeclampsia / HELLP Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Rasheedy Ali, principal investigator, Ain Shams University
Other Study IDs: ainshamHE4
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Human epididymis protein 4 — Human epididymis protein 4 serum level in predicting persistent proteniuria

SUMMARY:
Pre-eclampsia seems to be associated with a four to five times increase risk of later microalbuminuria and CKD which might suggest a possible direct renal damage from pre-eclampsia

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women 18-35 years old.
2. Fulfilling the criteria for diagnosis of sever preeclampsia.
3. Fulfilling the criteria for diagnosis of HELLP syndrome

Exclusion Criteria:

1. Diabetes mellitus
2. Preexisting renal disease.
3. Chronic hypertension
4. Rheumatologic diseases
5. Adnexal mass.

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: The diagnosis is made after 20 weeks of gestation in previously normotensive women who develop:
  * Systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥110 mmHg and proteinuria (with or without signs and symptoms of significant end-organ dysfunction).
  * Systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg (with or without proteinuria) and one or more of the following signs and symptoms of significant end-organ dysfunction
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
protein in urine | 12 weeks postpartum
  proteinuria > 0.3 mg protein / mg creatinine.

IPD SHARING:
Plan to Share IPD: No